CLINICAL TRIAL: NCT05276934
Title: Prospective Assessment of Brain Imaging After Aneurysmal of AVM-related Intracranial Hemorrhage
Brief Title: Brain Imaging After Non-traumatic Intracranial Hemorrhage (SAVEBRAINPWI)
Acronym: SAVEBRAINPWI
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2021298
Record Dates: First submitted 2022-02-15; First posted 2022-03-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Aneurysm, Ruptured; Aneurysmal Subarachnoid Hemorrhage; Arteriovenous Malformations; Intracranial Aneurysm; Intracranial Hemorrhages
MeSH Terms: conditions — Aneurysm, Ruptured; Subarachnoid Hemorrhage; Arteriovenous Malformations; Intracranial Aneurysm; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evolution of brain imaging in Non-traumatic Intracranial Hemorrhage: This study will use an established local protocol for DCI and intracranial arterial vasospastic stenosis screening, and follow-up to make sure that all patients have the same protocol and don't lose any chance of improvement and good outcome
  Interventions: Diagnostic Test: Brain computed tomography

INTERVENTIONS:
Diagnostic Test: Brain computed tomography — This study will use an established local protocol for DCI and intracranial arterial vasospastic stenosis screening, and follow-up to make sure that all patients have the same protocol and don't lose any chance of improvement and good outcome : CT perfusion at different time intervals

SUMMARY:
The study is an observational prospective evaluation of an approved and unchanged clinical management, evaluating different diagnosis methods to assess brain perfusion in patients with an aneurysmal or AVM-related intracranial hemorrhage

DETAILED DESCRIPTION:
The study is a prospective description and evaluation of an approved and unchanged clinical management, evaluating already used different diagnosis methods to assess brain perfusion in patients with atraumatic (aneurysmal, AVM-related, unknown cause) intracranial hemorrhage.

ELIGIBILITY:
i. Inclusion Criteria

1. Age ≥ 18 years
2. Non-traumatic intracranial hemorrhage (subarachnoid hemorrhage secondary to a ruptured aneurysm or AVM, unknown cause, per procedural bleed)
3. In case of ruptured aneurysm, AVM or other etiology : need to be secured with surgical clipping or endovascular intervention if judged possible
4. No contra-indication to perfusion imaging
5. Subject or legal representative is able and willing to give informed consent.

ii. Exclusion Criteria

1. Traumatic intracranial hemorrhage
2. Contra-indication to imaging or patient's refusal.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fit the inclusion criteria (suffered a non-traumatic (aneurysmal, AVM-related, unknown cause) intracranial hemorrhage) will be included prospectively.
  The deadline for data collection November, 2031 Data analysis will be performed when judged necessary by the investigators.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in brain hypoperfusion | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion Time to drain (seconds) on CT and/or MR perfusion

SECONDARY OUTCOMES:
Change in vessel size | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Change in the vessel size measured on digital subtraction angiography (DSA) and computed tomography angiogram (CTA) in millimeters
Time to next endovascular intervention for vasospastic stenosis | Number of days after the endovascular procedure until the next procedure in days, up to 4 weeks
  Delay between two procedures for the same indication
Transcranial Doppler | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Reduction in intracranial vasospasm assessed by the targeted vessel velocity in meters per second
Brain Hypoperfusion 2 | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Reduction in brain hypoperfusion assessed by the volumes on different perfusion parameters time to peak (in seconds) on CT and/or MR perfusion
Change in Glasgow coma scale | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Glasgow coma scale (GCS between 3 and 15, a higher score means a better outcome)
Change in National Institutes of Health Stroke Scale score | Change between day 0, 5, 9 after Intracranial Hemorrhage
  National Institutes of Health Stroke Scale (NIHSS between 0 and 42, a higher score means a worse outcome)
Change in the monitoring of tissue oxygen pressure (PtiO2) | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Monitoring of tissue oxygen pressure (PtiO2)
Change in the number of new ischemic lesions | Change between day 0, 5, 9, 21 after Intracranial Hemorrhage
  Number of new ischemic lesions on non-contrast CT scan
modified Rankin Scale at 3 months | 3 months after Intracranial Hemorrhage
  clinical evolution (mRS between 0 and 6, a higher score means a worse outcome)
Change in brain hypoperfusion 3 | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion parameters TMax maps in seconds on CT and/or MR perfusion
Change in brain hypoperfusion 4 | Change between day 0, 5, 9 after Intracranial Hemorrhage
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion parameters Mean transit time on CT and/or MR perfusion in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Guenego, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
No data sharing